CLINICAL TRIAL: NCT01905917
Title: The Singapore Tele-technology Aided Rehabilitation in Stroke (STARS) Study: A Randomized Controlled Trial
Brief Title: The Singapore Tele-technology Aided Rehabilitation in Stroke (STARS) Study
Acronym: STARS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: Singapore Millennium Foundation (Unknown); Singapore General Hospital (Other); Ang Mo Kio - Thye Hua Kwan Hospital (Other)
Responsible Party: Principal Investigator, Gerald Koh, Associate Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: The STARS Study
Record Dates: First submitted 2013-07-18; First posted 2013-07-23 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Stroke
Keywords: Stroke
MeSH Terms: conditions — Stroke | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Usual care
- Tele-Rehabilitation (Experimental): A tele-rehabilitation intervention involving weekly video-conferencing with a therapist, training exercise videos and use of wearable sensors to capture patient participation in exercises.
  Interventions: Other: Tele-rehabilitation

INTERVENTIONS:
Other: Tele-rehabilitation
  Arms: Tele-Rehabilitation

SUMMARY:
The primary hypothesis tested in this randomized control trial is that a tele-rehabilitation intervention involving video-conferencing with a therapist and use of wearable monitoring devices in the first three months after stroke results greater functional recovery using the Jette Late Life Functional and Disability Instrument (LLFDI) (primary outcome) among stroke at three months survivors compared to usual care.

The secondary hypotheses tested in this randomized control trial are that a tele-rehabilitation intervention involving video-conferencing with a therapist and use of wearable monitoring devices in the first three months after stroke results in:

* Functional recovery using the LLFDI at 6 months,
* Functional recovery using gait speed, 2-minute walk test and Shah modified Barthel Index at 3 and 6 months,
* Greater contact time with a therapist at 3 & 6 months,
* Better balance at 3 & 6 months,
* Better self-report health-related quality of life at 3 & 6 months,
* Decreased health service utilization at 3 & 6 months,
* Reduced caregiver burden at three months survivors compared to usual care at 3 & 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 40 years;
2. Recent stroke (defined as stroke symptoms occurring within 4 weeks prior to admission into community hospitals);
3. Diagnosis of stroke made by clinician and/or supported by brain imaging;
4. Able to sit unsupported for 30 seconds;
5. Able to stand on the non-paretic leg for >4 sec;
6. Able to walk at least 2m with maximum of 1 person assist;
7. Able to follow a 3-step command;
8. Living in the community before discharge and expected to be discharged home;
9. Has a caregiver.

Exclusion Criteria:

1. Has a pacemaker in-situ (because of possible interference of pacemakers by wireless electronic signals);
2. Unable to ambulate at least 150 feet prior to stroke, or intermittent claudication while walking less than 200 meters;
3. Serious cardiac conditions (hospitalization for myocardial infarction or heart surgery within 3 months, history of severe congestive heart failure, serious and unstable cardiac arrhythmias, hypertrophic cardiomyopathy, severe aortic stenosis, angina or dyspnea at rest or during activities of daily living);
4. History of serious chronic obstructive pulmonary disease or oxygen dependence;
5. Severe weight bearing pain;
6. Pre-existing neurological disorders such as Parkinson's disease, Amyotrophic Lateral Sclerosis (ALS), Multiple Sclerosis (MS) or severe dementia
7. History of major head trauma with severe residual deficits;
8. Lower extremity amputation;
9. Legal blindness or severe visual impairment;
10. Severe uncontrolled psychiatric illness such as psychosis, schizophrenia or medication refractory depression;
11. Life expectancy less than three months;
12. Severe arthritis or orthopedic problems that limit passive ranges of motion of lower extremity (knee flexion contracture of > 10°, knee flexion ROM < 90°, hip flexion contracture > 25°, and ankle plantar flexion contracture > 15°);
13. History of sustained alcoholism or drug abuse in the last six months;
14. Hypertension with systolic blood pressure greater than 200 mmHg and diastolic blood pressure greater than 110 mmHg at rest, that cannot be medically controlled into the resting range of 180/100 mmHg.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2013-11; Primary Completion 2017-03 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Jette Late Life Functional and Disability Instrument (LLFDI) | 3 months
  Disability component of the Jette Late Life Functional and Disability Instrument (LLFDI)

SECONDARY OUTCOMES:
Jette Late Life Functional and Disability Instrument (LLFDI) | 6 months
  Disabiity component of Jette Late Life Functional and Disability Instrument (LLFDI)

OTHER OUTCOMES:
Gait speed | 3 & 6 months
  Gait speed
Two-Minute Walk test | 3 & 6 months
  Two-Minute Walk test
Shah-modified Barthel Index | 3 & 6 months
  Shah-modified Barthel Index
Activities-Specific Balance Confidence Scale | 3 & 6 months
  Activities-Specific Balance Confidence Scale
Self-reported health-related quality-of-life using the Euro-QOL (EQ-5D) | 3 & 6 months
  Self-reported health-related quality-of-life using the Euro-QOL (EQ-5D)
Health service utilization (perform cost-effectiveness analyses) using the Singapore Stroke Study Health Service Utilization Form | 3 & 6 months
  Health service utilization (perform cost-effectiveness analyses) using the Singapore Stroke Study Health Service Utilization Form
Caregiver reported stress using the Zarit Caregiver Burden Inventory | 3 & 6 months
  Caregiver reported stress using the Zarit Caregiver Burden Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Cheng Yes, PhD, Principal Investigator — National University of Singapore; Tay Arthur, PhD, Principal Investigator — National University of Singapore
Locations (2):
- Singapore (2):
  - Singapore General Hospital, Singapore
  - Ang Mo Kio Thye Hua Kwan Hospital, Singapore

REFERENCES:
- [Background] Duncan PW, Sullivan KJ, Behrman AL, Azen SP, Wu SS, Nadeau SE, Dobkin BH, Rose DK, Tilson JK, Cen S, Hayden SK; LEAPS Investigative Team. Body-weight-supported treadmill rehabilitation after stroke. N Engl J Med. 2011 May 26;364(21):2026-36. doi: 10.1056/NEJMoa1010790. PMID 21612471
- [Background] Duncan PW, Sullivan KJ, Behrman AL, Azen SP, Wu SS, Nadeau SE, Dobkin BH, Rose DK, Tilson JK; LEAPS Investigative Team. Protocol for the Locomotor Experience Applied Post-stroke (LEAPS) trial: a randomized controlled trial. BMC Neurol. 2007 Nov 8;7:39. doi: 10.1186/1471-2377-7-39. PMID 17996052
- [Background] Chumbler NR, Quigley P, Li X, Morey M, Rose D, Sanford J, Griffiths P, Hoenig H. Effects of telerehabilitation on physical function and disability for stroke patients: a randomized, controlled trial. Stroke. 2012 Aug;43(8):2168-74. doi: 10.1161/STROKEAHA.111.646943. Epub 2012 May 24. PMID 22627983
- [Derived] Koh GC, Yen SC, Tay A, Cheong A, Ng YS, De Silva DA, Png C, Caves K, Koh K, Kumar Y, Phan SW, Tai BC, Chen C, Chew E, Chao Z, Chua CE, Koh YS, Hoenig H. Singapore Tele-technology Aided Rehabilitation in Stroke (STARS) trial: protocol of a randomized clinical trial on tele-rehabilitation for stroke patients. BMC Neurol. 2015 Sep 5;15:161. doi: 10.1186/s12883-015-0420-3. PMID 26341358
- See also: Singapore Millennium Foundation — http://www.smf-scholar.org/